CLINICAL TRIAL: NCT06444386
Title: Electrocardiographic Imaging of MultiPoint Pacing and SyncAV: Understanding Optimized Programming for Cardiac Resynchronization Therapy
Brief Title: ECGi of SyncAV With MultiPoint Pacing
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10292
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MPP + SyncAV — Cardiac resynchronization therapy (CRT) features of MultiPoint Pacing (MPP) and SyncAV (dynamic atrioventricular delay programming) enabled.

SUMMARY:
The objective of this clinical study was to evaluate the impact of Multipoint Pacing (MPP) and SyncAV programming on ventricular electrical activation time and activation sequence using noninvasive electrocardiographic imaging (ECGi) in patients receiving cardiac resynchronization therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients previously implanted with a SyncAV and MPP-enabled Abbott Quadripolar CRT pacing system
* Patient must be > 18 years of age, able to provide informed consent and willing to comply with study requirements
* Sinus (or atrial paced) rhythm with intact AV conduction with PR interval ≤ 250 ms
* Patient has documented Left Bundle Branch Block (LBBB)

Exclusion Criteria:

* Resting heart rate > 100 bpm
* AV Block (1st degree with PR> 250 ms, 2nd or 3rd degree)
* Documented persistent atrial tachycardia or atrial fibrillation at the moment of enrollment or patients not likely to remain in sinus (or atrial paced) rhythm for the duration of the study
* Recent (< 3 months) myocardial infarction, ablation, electrolyte imbalance, or any condition within the last 90 days that would contraindicate for CRT programming changes in the opinion of the investigator
* Women who are pregnant or plan to become pregnant during the study course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population for this clinical investigation consisted of patients over the age of 18 years who have been previously implanted with an Abbott CRT device capable of SyncAV and MultiPoint Pacing. This clinical investigation enrolled male and female subjects from the general heart failure population. Subjects must have met all eligibility criteria and provide written informed consent prior to conducting any investigation-specific procedures not considered standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Left ventricular activation time | 1 day
  Evaluate acute changes in left ventricular (LV) electrical activation time measured with ECGi resulting from various CRT pacing configurations with MPP and SyncAV

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No